CLINICAL TRIAL: NCT05322447
Title: Effect of High-dose L-Carnitine Supplementation on Diaphragmatic Function Assessed by Ultrasonography in Critically Ill Patients With Respiratory Failure: a Randomized Clinical Trial
Brief Title: High-dose L-Carnitine and Diaphragmatic Function Assessed by Ultrasonography in Patients With Respiratory Failure.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R / 2022
Record Dates: First submitted 2022-03-21; First posted 2022-04-11 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): maintenance dose of L- carnitine 6 gm/day to keep normal level (normal L-carnitine level is normal 25-50 mmol/L)
  Interventions: Drug: L Carnitine ( low dose)
- experimental group (Experimental): high dose of L- Carnitine 18 gm/day as a continuous intravenous infusion to reach double the normal plasma level.
  Interventions: Drug: L-Carnitine ( high dose)

INTERVENTIONS:
Drug: L Carnitine ( low dose) — will receive a maintenance dose of L- carnitine 6 gm/day to keep normal level (normal L-carnitine level is normal 25-50 mmol/L)
  Arms: Control Group
Drug: L-Carnitine ( high dose) — will receive a high dose of L- Carnitine 18 gm/day as a continuous intravenous infusion to reach double the normal plasma level
  Arms: experimental group

SUMMARY:
L-Carnitine supplementation has been shown to boost muscular performance in several studies. In hemodialysis patients with muscular weakness, fatigue, or cramps/aches, after L-carnitine treatment, about two-thirds of patients had at least some improvement in muscular symptoms . L-Carnitine was also found to improve the left ventricular ejection fraction (LVEF) in hemodialysis patients with cardiac morbidity who had significantly reduced LVEF in echocardiography before supplementation. Moreover, L-Carnitine has been shown to improve muscular function and exercise performance in athletes in several studies

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 years old or greater
* Both genders have respiratory failure either of the primary medical origin or in the post-surgical course.
* Not in need of mechanical ventilation

Exclusion Criteria:

* Renal failure on regular dialysis
* Hypothyroidism
* Seizures
* End-stage liver disease
* Mechanical ventilation
* History or discovered allergy to L-carnitine, pivampicillin, and other pivalate-conjugated antibiotics.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound diaphragmatic function | at days 7
  Diaphragmatic excursion by ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, Cairo
  - Mona A Ammar, Cairo